CLINICAL TRIAL: NCT06357845
Title: Healthy Futures Research Study: Linking Somatic Mutation Rate With Baseline Exposure in East Palestine
Brief Title: Linking Somatic Mutation Rate With Baseline Exposure in East Palestine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CASE5Z24; 1R21ES036031-01 (NIH)
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Somatic Mutation
Keywords: East Palestine; Train Derailment; Healthy Futures Research Study; Environmental Impact
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: A cross-sectional study design will be implemented.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Residents effected by the Derailment event (Other): Eligible residents must be adult participants from Columbiana County, Ohio, Mahoning County, Ohio, Beaver County, Pennsylvania, or Lawrence County, Pennsylvania.
  Interventions: Other: Survey; Other: Biological specimen collection; Other: Communications about study updates and future research opportunities; Other: Qualitative interview

INTERVENTIONS:
Other: Survey — Participants will complete a brief web-based survey asking about their experiences related to the February 3, 2023 train derailment, health experiences and concerns following the derailment, and background information regarding their health history. The survey will last approximately 15 minutes.
Other: Biological specimen collection — Participants may possibly contribute biospecimens such as blood, spit, hair, and/or toenail clippings. Participants will be asked which samples they are interested in providing. Participants will receive a specific sample collection kit based on their selection. For blood samples, participants will receive a mailed collection kit at their mailing address. A member of the research team will reach out to schedule blood sample collection, which may take place at home with a trained phlebotomist or at a designated collection site. A total of 1-2 teaspoons of blood (5-10 milliliters) will be collected at a one-time blood draw. For either saliva, hair, and/or toenail clippings, participants will be sent a sample collection kit and receive instructions at their mailing address. This kit also includes a return mailing envelope. Participants will provide the selected samples in the collection kits, place them in the return mailing envelope, and send them back to the research team.
Other: Communications about study updates and future research opportunities — By consenting to participate in this study, the research team will send updates about the research results and any additional study opportunities to participants.
Other: Qualitative interview — A total of 40 study participants will be recruited to participate in a 90-minute interview with open-ended questions. The interviews will be video and audio-recorded.

SUMMARY:
The goal of this study is to This research team is conducting this study to develop methods to measure the biological impact of exposure to the chemicals released following the February 3, 2023 train derailment on residents of East Palestine, Ohio, and surrounding communities. The main question it aims to answer is:

* What biological impact will be measured based on DNA damage?
* In participants who provide a biospecimen, how are biomarker changes related to proximity to the derailment and variations in residents' health histories and behaviors?

Participants will:

* Complete a brief survey asking about experiences related to the February 3, 2023 train derailment, health experiences, and concerns following the derailment, and background information regarding health history.
* Possibly contribute biospecimens such as blood, spit, hair, and/or toenail clippings.
* Receive communication about study updates and future research opportunities.
* A total of 40 study participants will be recruited to participate in a 90-minute interview. The interviews will be video and audio recorded.

DETAILED DESCRIPTION:
On February 3, 2023, at 8:55 pm EST, over 30 train cars from a Norfolk Southern train carrying hazardous chemicals derailed in the village of East Palestine, Ohio. In a few hours, residents within a 1- mile radius were ordered to evacuate, followed by several shelter-in-place orders. By February 6, the evacuation zone was expanded, and a controlled burn was implemented in the hopes of preventing an explosion. A week later, the Environmental Protection Agency (EPA) announced vinyl chloride, butyl acrylate, ethylhexyl acrylate, and ethylene glycol monobutyl ether were released into the air, surface soil, and surface waters. Although the EPA failed to detect contaminants at concerning levels for human health in the East Palestine region on February 12, East Palestine residents with private wells were recommended to use bottled water only four days later, and subsequent testing has detected elevated chemical levels in the region. The EPA instructed Norfolk Southern to expand testing and include dioxin testing on March 2. Four days later seven members of a 15-person CDC/ATSDR team reported sore throats, headaches, coughing and nausea after conducting Assessment of Chemical Exposure (ACE) surveys. The inconsistent messaging from the EPA and other governmental agencies have frustrated East Palestine and surrounding community (EPSC) residents, and generated concerns regarding long-term health effects.

This study has several aims:

* Establish the Healthy Futures Pilot Cohort utilizing a community-engaged research approach
* Compare genotoxicity levels arising from chemical exposure by geographical proximity and direction from the train derailment epicenter utilizing the somatic mutation rate in DNA among residents
* Understand experiences during and post-disaster with respect to effects on quality of life, perceived stressors, future prospects, and overall health-and how acute disasters shape risk perception, coping strategies, and access to health-protective resources through semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Residence on February 3rd, 2023 in Columbiana County, Ohio, Mahoning County, Ohio, Beaver County, PA, or Lawrence County, PA.
* Current residence in the United States.

Exclusion Criteria:

* Address provided for February 3rd, 2023 not in Columbiana County, Ohio, Mahoning County, Ohio, Beaver County, PA, or Lawrence County, PA
* Invalid address provided for February 3rd, 2023 residence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Geographic Association of Somatic Mutation Rates | Up to 24 months
  The primary outcome measure is somatic mutation rates in association with geographical distance from the train derailment epicenter.

SECONDARY OUTCOMES:
Self-reported Symptomology Association of Somatic Mutation Rates | Up to 24 months
  The secondary outcome measure is somatic mutation rates in association with self-reported symptomology at time of exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick R Schumacher, PhD, Principal Investigator — Case Western Reserve University, Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Questionnaire data will be captured by usage of REDCap and Qualtrix data bases. Genomic data, low pass sequencing measuring the somatic mutation rate (SMR), will be individual level data.
Time Frame: Genomic data will be uploaded to dbGAP within three months of data generation and released within six months to individuals with approved protocols.
Access Criteria: Submitted proposal and approved by the study data access committee. All proposals need to be related to the primary and secondary hypotheses.
URL: https://www.ncbi.nlm.nih.gov/gap/